CLINICAL TRIAL: NCT05601401
Title: Phase II Clinical Study to Assess the Efficacy and Safety of Recombinant Humanized Anti-HER2 Monoclonal Antibody MMAE Coupling Agent in Treating Patients With Locally Advanced or Metastatic Salivary Gland Tumors Expressing HER2
Brief Title: Phase II Study of RC48-ADC in Treating Patients With Salivary Gland Tumors Expressing HER2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RCVDORIIR002
Record Dates: First submitted 2022-10-17; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Salivary Gland Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm (Experimental): Patients receive RC48-ADC.
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC — RC48-ADC 2.0 mg/kg IV every 14 days
  Other Names: RC48

SUMMARY:
The goal of this clinical trial is to learn about the efficacy and safety of RC48-ADC, a HER2-targeting antibody-drug conjugate, in patients with HER2-positive and HER2-low expressing advanced or metastatic salivary cancer.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the efficacy and safety of RC48-ADC, a HER2-targeting antibody-drug conjugate, in patients with HER2-positive and HER2-low expressing advanced or metastatic salivary cancer. Participants will receive RC48-ADC 2.0 mg/kg intravenous (IV) infusion each 14-day treatment cycle until disease progression (PD) (as assessed by the investigator), unmanageable toxicity, or study termination.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent to participate in the research and sign the informed consent form;
2. Male or female, age ≥ 18;
3. Expected survival time ≥ 12 weeks;
4. Locally advanced or metastatic salivary gland malignant tumor confirmed by histopathology that cannot be completely resected by surgery;
5. Subjects who have not received systemic anti-tumor treatment after being diagnosed as locally advanced or metastatic salivary gland malignant tumor that cannot be removed surgically; Or disease progression occurs after receiving at least first-line systematic treatment in the past, in which the patient has disease progression within 12 months after receiving neoadjuvant or adjuvant chemotherapy, and can be included in this clinical study;
6. Have measurable lesions specified in RECIST v1.1 standard;
7. Subjects can provide the primary or metastatic tumor samples for HER2 detection; HER2 IHC is 2+or 3+;
8. ECOG physical condition score 0-2;
9. Adequate heart, bone marrow, liver and kidney functions (subject to the normal value of the research center):

   * ① Left ventricular ejection fraction ≥ 50%;
   * ② Hemoglobin ≥ 9g/dL;
   * ③ Absolute neutrophil count (ANC) ≥ 1.5 × 109/L；
   * ④ Platelet ≥ 100 × 109/L；
   * ⑤ In patients without liver metastasis, serum total bilirubin ≤ 1.5 times the upper limit of normal value (ULN); Total serum bilirubin in patients with liver metastasis ≤ 3 × ULN；
   * ⑥ ALT and AST ≤ 2.5 in the absence of liver metastasis × ULN, ALT and AST ≤ 5 in case of liver metastasis × ULN；
   * ⑦ Blood creatinine ≤ 1.5 × ULN；
10. For female subjects: they should be surgical sterilized or postmenopausal patients, or agree to use at least one medically approved contraceptive measure (such as intrauterine device [IUD], contraceptives or condoms) during the study treatment period and within 6 months after the end of the study treatment period. The serum or urine pregnancy test must be negative within 7 days before the study enrollment, and they must be non lactating. Male subjects should agree to use at least one medically approved contraceptive measure (such as condom, abstinence, etc.) during the study treatment period and within 6 months after the end of the study treatment period;
11. Willing and able to follow the trial and follow-up procedures.

Exclusion Criteria:

1. Known allergic to recombinant humanized anti HER2 monoclonal antibody MMAE coupling agent drugs and their related components;
2. Have received anti-tumor treatment (including chemotherapy, radiotherapy, immunotherapy, etc.) or participated in other clinical research treatments within 3 weeks before the start of the study treatment, or the toxicity related to the previous anti-tumor treatment has not recovered to grade 0-1 (except grade 2 alopecia);
3. He has been treated with recombinant humanized anti HER2 monoclonal antibody MMAE coupling agent in the past;
4. Major surgery was carried out within 4 weeks before the start of the study drug administration and it was not completely recovered;
5. Other serious and uncontrollable concomitant diseases that may affect the protocol compliance or interfere with the interpretation of results, including active infection or progressive (serious) infection, uncontrollable diabetes Cardio cerebral vascular disease (Grade III or IV heart failure defined by New York Heart Association, more than Grade II heart block, acute myocardial infarction, unstable arrhythmia or unstable angina pectoris in the past 6 months, cerebral infarction in the past 6 months, except lacunar cerebral infarction) or pulmonary disease (interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm history), deep vein thrombosis or pulmonary embolism;
6. Patients with other malignant tumors within 3 years before the start of the study drug administration, but excluding obviously cured malignant tumors or curable cancers, such as basal skin cancer or squamous cell skin cancer, localized low-risk prostate cancer, cervical carcinoma in situ or breast carcinoma in situ; Remarks: Limited low-risk prostate cancer (defined as patients with stage ≤ T2a, Gleason score ≤ 6 and PSA<10ng/mL (if measured) at the time of diagnosis of prostate cancer who have received radical treatment and have no biochemical recurrence of prostate specific antigen (PSA) can participate in this study);
7. Have central nervous system (CNS) metastasis and/or cancerous meningitis. Subjects who have received brain metastasis treatment can consider participating in this study, provided that the condition is stable for at least 3 months, no disease progression is confirmed by imaging examination within 4 weeks before the first administration of the study, and all neurological symptoms have recovered to the baseline level, there is no evidence that new or expanded brain metastasis has occurred, and radiation, surgery or steroid treatment is stopped at least 28 days before the first administration of the study treatment. This exception does not include malignant meningitis, regardless of its clinical stability should be excluded;
8. Pregnant or lactating women;
9. HIV test result is positive;
10. Patients with active hepatitis B or hepatitis C

    * ① HBsAg positive persons also detected positive copy number of HBV DNA; HBV DNA must be detected when such patients are studied and screened;
    * ② Patients with positive HCV antibody test results can only be included in this study if the PCR test result of HCV RNA is negative.
11. There are active or progressive infections requiring systematic treatment, such as active pulmonary tuberculosis;
12. Suffering from any other disease, metabolic abnormality, physical examination abnormality or laboratory examination abnormality, according to the judgment of the investigator, it is reasonable to suspect that the patient has a certain disease or state that is not suitable for the use of the study drug, or will affect the interpretation of the study results, or put the patient at high risk;
13. It is estimated that the patient's compliance to participate in this clinical study is insufficient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first. Assessed up to 24 months.
  Tumor response was assessed by investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Objective Response Rate （ORR） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first. Assessed up to 24 months.
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR).
Overall Survival (OS) | From date of randomization until the date of death from any cause. Assessed up to 60 months.
  OS was defined as the time from the date of randomization to the date of death from any cause.
Disease Control Rate （DCR） | Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first. Assessed up to 60 months.
  CR+PR+SD

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No